CLINICAL TRIAL: NCT06499753
Title: Differences in Dry Eye Symptoms Related to Geographic Location in Spain and Impact of Artificial Tears Use
Acronym: EMO-01
Status: Completed | Type: Observational
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Raul Martin Herranz, PhD, University of Valladolid
Other Study IDs: UVaGiO-PI201606
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Syndromes; Hyaluronic Acid; OSDI
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: high molecular weight HA-based artificial tears — use of high molecular weight HA-based artificial tears three times per day

SUMMARY:
This study assessed the differences in DED symptomatology measured with the OSDI questionnaire regarding climate data of the geographic location in a large population in Spain, with a special focus on the relative humidity (RH) of the place of residence and the impact of artificial tears use, to help eye care practitioners in patient management and education

DETAILED DESCRIPTION:
This was a multicentre study enrolling patients to attend primary eye care centres of the EMO research group across 12 different Spanish locations. A comprehensive eye examination was performed in all participants. Dryness symptomatology was assessed with OSDI questionnaire. In subjects with dryness symptomatology (OSDI questionnaire score between 13 and 32) were prescribed to use high molecular weight HA-based artificial tears (DISOP Inc, Spain) along three months), instilled 3 times per day.

Additionally, the daily mean, minimum, and maximum values of the climate data for five different variables [skin temperature (°C), wind gusts (m/s), air temperature (°C), atmospheric pressure (Pa) and RH (%)] corresponding to the visit date were collected from the EU-funded Copernicus Climate Change Service and the 5-year average RH values published by the Spanish meteorological agency.

ELIGIBILITY:
Inclusion Criteria:

• Volunteer subjects of legal age will be included who agree to participate in the study after being informed by the researcher of each center

Exclusion Criteria:

* Hyperthyroidis
* Rheumatism
* Lupus
* Autoimmune disease
* Previous diagnosis of Dye Eye Disease
* Cicatricial conjunctivitis
* Pterygium
* Eyelid trichiasis
* History of any eye medication use in the last 3 months to treat any eye condition (glaucoma, etc.)
* Active anterior eye inflammation (such as blepharitis, conjunctivitis, keratitis, scleritis, uveitis, etc.)
* Use of contact lenses in the last 3 months
* Previous ocular trauma or surgery in the last 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
OSDI Score | three months
  Change in the Ocular Surface Disease Index (OSDI) score ranged from 0 (asymptomatic) to 100 (severe dry eye)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Martin, PhD, Principal Investigator — IOBA Eye Institute
Locations (1):
- IOBA Eye Institute, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be available by request to PI